CLINICAL TRIAL: NCT00339235
Title: Establishment of a Clinical Perinatal Database and Bank of Biological Materials
Brief Title: Establishment of a Perinatal Database and a Bank of Biological Materials
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998001; OH98-CH-N001
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Labor; Preterm Birth; Pregnancy
Keywords: Preterm Birth Prevention; Preterm Birth; Pregnancy; Pregnancy Complications; Natural History
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Non-pregnant women: Non-pregnant women aged 18 years and older
- Pregant women: Pregnant women aged 18 years and older

SUMMARY:
The aim of this project is to establish a clinical database and a bank of biological materials which will be used to improve the pathophysiologic understanding of the mechanisms underlying various pregnancy diseases. The US-Mexico Reproductive Health Research Development Workshop, sponsored by the NIH, recommended that the setting up of "tissue, blood, and placental banks from human and relevant animal models should be developed to aid in understanding how prenatal conditions relate to pathological consequences in adult life".

A large observational study in the United States of America, the National Collaborative Perinatal Project (NCPP), was conducted over 30 years ago (1959-1966) and has yielded a large amount of useful information. However standards of obstetrical and neonatal care have changed significantly over the last 30 years. Thus the setting up of a contemporary clinical perinatal database and bank of biological materials is required. In order to obtain sufficient data for statistical analysis a large sample size is necessary.

We propose to carry out this project at Sotero del Rio Hospital, Santiago Chile as this hospital has a delivery rate of approximately 14,000 women per year. Previous research collaborative efforts between the Sotero del Rio Hospital and the PRB have been carried out in compliance with NIH research regulations. Sotero del Rio Hospital has had previous successful negotiations of Single Project Assurances (SPA) with the NIH.

Information will be collected from clinical history taking, physical examination, sonographic examination and standard laboratory procedures. The bank of biological fluids and tissues will include maternal blood, umbilical cord plasma, amniotic fluid, maternal urine and placental tissue. No procedures will be carried out on patients that are not part of standard of care at Sotero del Rio Hospital.

DETAILED DESCRIPTION:
The aim of this project is to establish a clinical database and a bank of biological materials which will be used to improve the pathophysiologic understanding of the mechanisms underlying various pregnancy diseases. The US-Mexico Reproductive Health Research Development Workshop, sponsored by the NIH, recommended that the setting up of "tissue, blood, and placental banks from human and relevant animal models should be developed to aid in understanding how prenatal conditions relate to pathological consequences in adult life".

A large observational study in the United States of America, the National Collaborative Perinatal Project (NCPP), was conducted over 30 years ago (1959-1966) and has yielded a large amount of useful information. However standards of obstetrical and neonatal care have changed significantly over the last 30 years. Thus the setting up of a contemporary clinical perinatal database and bank of biological materials is required. In order to obtain sufficient data for statistical analysis a large sample size is necessary.

We propose to carry out this project at Sotero del Rio Hospital, Santiago Chile as this hospital has a delivery rate of approximately 14,000 women per year. Previous research collaborative efforts between the Sotero del Rio Hospital and the PRB have been carried out in compliance with NIH research regulations. Sotero del Rio Hospital has had previous successful negotiations of Single Project Assurances (SPA) with the NIH.

Information will be collected from clinical history taking, physical examination, sonographic examination and standard laboratory procedures. The bank of biological fluids and tissues will include maternal blood, umbilical cord plasma, amniotic fluid, maternal urine and placental tissue. No procedures will be carried out on patients that are not part of standard of care at Sotero del Rio Hospital.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Women who receive care at participating units will be eligible for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending Detroit Medical Center (DMC) prenatal clinics in Detroit.Non-pregnant women attending DMC clinics are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 30570 (Actual)
Dates: Start 1998-01-06; Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
1.Maternal mortality 2.Route of delivery 3.Infection related complications 4.Bleeding, blood loss and transfusion requirements 5.Hypertensive disorders 6.Venous and arterial thrombotic events 7. Any other complications of pregnancy, labor or del... | Ongoing
  Data and specimen analysis is ongoing

SECONDARY OUTCOMES:
Birthweight; Perinatal mortality; Congenital anomalies; Intrauterine growth retardation; Respiratory distress syndrome; Chronic pulmonary disease; Intraventricular hemorrhage;Necrotizing enterocolitis; Retinopathy of prematurity | Ongoing
  Birthweight; Perinatal mortality; Congenital anomalies; Intrauterine growth retardation; Respiratory distress syndrome; Chronic pulmonary disease; Intraventricular hemorrhage;Necrotizing enterocolitis; Retinopathy of prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Wilkins-Haug L, Roberts DJ, Morton CC. Confined placental mosaicism and intrauterine growth retardation: a case-control analysis of placentas at delivery. Am J Obstet Gynecol. 1995 Jan;172(1 Pt 1):44-50. doi: 10.1016/0002-9378(95)90082-9. PMID 7847559
- [Background] Pollack RN, Divon MY. Intrauterine growth retardation: definition, classification, and etiology. Clin Obstet Gynecol. 1992 Mar;35(1):99-107. doi: 10.1097/00003081-199203000-00015. No abstract available. PMID 1544253
- [Background] Branch DW, Andres R, Digre KB, Rote NS, Scott JR. The association of antiphospholipid antibodies with severe preeclampsia. Obstet Gynecol. 1989 Apr;73(4):541-5. PMID 2494618